CLINICAL TRIAL: NCT02854319
Title: REPRISE EDGE: REpositionable Percutaneous Replacement of NatIve StEnotic Aortic Valve Through Implantation of LOTUS EDGE Valve System - Evaluation of Performance and Safety
Brief Title: REpositionable Percutaneous Replacement of NatIve StEnotic Aortic Valve Through Implantation of LOTUS EDGE Valve System
Acronym: REPRISE EDGE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigational Medical Device is not available and the 15 patients enrolled completed their 1-yr follow-up per protocol
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S2367
Record Dates: First submitted 2016-07-28; First posted 2016-08-03 (Estimated); Last update posted 2018-05-31 (Actual); Status verified 2018-05

CONDITIONS: Aortic Valve Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LOTUS Edge Valve System (Experimental): Transcatheter aortic valve implantation (TAVI) with the LOTUS Edge™ Valve System when used with the Lotus™ or iSleeve™ Introducer Set
  Interventions: Device: LOTUS Edge Valve System

INTERVENTIONS:
Device: LOTUS Edge Valve System — Transcatheter Aortic Valve Implantation (TAVI) with the LOTUS Edge™ Valve System when used with the Lotus™ or iSleeve™ Introducer Set

SUMMARY:
The objective of the REPRISE EDGE study is to confirm the acute performance and safety of the LOTUS Edge™ Valve System when used with the Lotus™ or iSleeve™ Introducer Set for transcatheter aortic valve implantation (TAVI) in symptomatic patients with severe calcific aortic stenosis who are considered high risk for surgical valve replacement.

DETAILED DESCRIPTION:
This clinical study is a prospective, single-arm study designed to demonstrate that the acute performance and safety of the LOTUS Edge Valve System when used with the iSleeve or Lotus Introducer Set are consistent with the results of the commercially approved Lotus Valve System used in the REPRISE II study, when delivered and deployed in symptomatic subjects who have severe calcific aortic valve stenosis and who are at high risk for surgical aortic valve replacement (SAVR).

ELIGIBILITY:
Inclusion Criteria:

1. Subject is ≥70 years of age.
2. Subject has documented calcific native aortic valve stenosis with an initial aortic valve area (AVA) of <1.0 cm2 (or AVA index of <0.6 cm2/m2) and either a mean pressure gradient >40 mm Hg or a jet velocity >4 m/s, as measured by echocardiography and/or invasive hemodynamics.

   Note: In cases of low flow, low gradient aortic stenosis dobutamine can be used to assess the grade of aortic stenosis (maximum dobutamine dose of 20 mcg/kg/min recommended)c; the subject may be enrolled if echocardiographic criteria are met with this augmentation.
3. Subject has a documented aortic annulus size between ≥20 mm and ≤27 mm based on pre-procedure diagnostic imaging.
4. Subject has symptomatic aortic valve stenosis with NYHA Functional Class ≥ II.
5. Subject is considered high risk for surgical valve replacement based on at least one of the following:

   * STS score ≥8%, and/or
   * Agreement by the heart team (which must include an in-person evaluation by an experienced cardiac surgeon) that subject is at high operative risk of serious morbidity or mortality with surgical valve replacement.
6. Heart team (which must include an experienced cardiac surgeon) assessment that the subject is likely to benefit from valve replacement
7. Subject (or legal representative) understands the study requirements and the treatment procedures, and provides written informed consent.
8. Subject, family member and/or legal representative agree(s) and subject is capable of returning to the study hospital for all required scheduled follow up visits.

Exclusion Criteria:

1. Subject has a congenital unicuspid or bicuspid aortic valve.
2. Subject with an acute myocardial infarction within 30 days of the index procedure (defined as Q-wave MI or non-Q-wave MI with total CK elevation ≥ twice normal in the presence of CK-MB elevation and/or troponin level elevation).
3. Subject has had a cerebrovascular accident or transient ischemic attack within the past 6 months, or has any permanent neurologic defect prior to study enrollment.
4. Subject is on dialysis or has serum creatinine level >3.0 mg/dL or 265 µml/L.
5. Subject has a pre-existing prosthetic aortic or mitral valve.
6. Subject has >3+ mitral regurgitation, >3+ aortic regurgitation or >3+ tricuspid regurgitation.
7. Subject has a need for emergency surgery for any reason.
8. Subject has a history of endocarditis within 12 months of index procedure or evidence of an active systemic infection or sepsis.
9. Subject has echocardiographic evidence of new intra-cardiac vegetation or intraventricular or paravalvular thrombus requiring intervention.
10. Subject has Hgb <9 g/dL, platelet count <50,000 cells/mm3 or >700,000 cells/mm3, or white blood cell count <1,000 cells/mm3.
11. Subject requires chronic anticoagulation therapy after the implant procedure and cannot be treated with warfarin (other anticoagulants are not permitted in the first month) for at least 1 month concomitant with either aspirin or clopidogrel.

    Note: An alternative P2Y12 inhibitor may be prescribed if subject is allergic to or intolerant of clopidogrel
12. Subject has had a gastrointestinal bleed requiring hospitalization or transfusion within the past 3 months, or has other clinically significant bleeding diathesis or coagulopathy that would preclude treatment with required antiplatelet regimen, or will refuse transfusions.
13. Subject has known hypersensitivity to contrast agents that cannot be adequately pre-medicated, or has known hypersensitivity to aspirin, all thienopyridines, heparin, nickel, titanium, or polyurethanes.
14. Subject has a life expectancy of less than 12 months due to non-cardiac, co-morbid conditions based on the assessment of the investigator at the time of enrollment.
15. Subject has hypertrophic obstructive cardiomyopathy.
16. Subject has any therapeutic invasive cardiac procedure within 30 days prior to the index procedure (except for balloon aortic valvuloplasty and pacemaker implantation which are allowed).
17. Subject has untreated coronary artery disease, which in the opinion of the treating physician, is clinically significant and requires revascularization.
18. Subject has documented left ventricular ejection fraction <30%.
19. Subject is in cardiogenic shock or has hemodynamic instability requiring inotropic support or mechanical support devices.
20. Subject has severe vascular disease that would preclude safe access (e.g., aneurysm with thrombus that cannot be crossed safely, marked tortuosity, significant narrowing of the abdominal aorta, severe unfolding of the thoracic aorta, or symptomatic carotid or vertebral disease).
21. Subject has arterial access that is not acceptable for the LOTUS Edge delivery system and its compatible Lotus or iSleeve Introducers as defined in the Directions For Use, or severe iliofemoral tortuosity or calcification that would prevent safe placement of either introducer sheath.
22. Current problems with substance abuse (e.g., alcohol, etc.).
23. Subject is participating in another investigational drug or device study that has not reached its primary endpoint.
24. Subject does not have a permanent pacemaker but has a class I or II indication for pacemaker implantation (based on the latest available ESC guidelines).

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-09-07 (Actual); Primary Completion 2016-10-25 (Actual); Study Completion 2018-03-13 (Actual)

PRIMARY OUTCOMES:
Mean aortic valve pressure gradient | At discharge from hospital or at 7 days post-procedure (whichever comes first)
  Mean aortic valve pressure gradient as measured by echocardiography and assessed by an independent core laboratory.

SECONDARY OUTCOMES:
Technical success | Immediately post-procedure (patient discharged from operative room)
  Defined as successful vascular access, delivery, and deployment of a Lotus Valve; successful retrieval with the delivery system; and correct positioning of a single Lotus Valve in the proper anatomical location (reported as percent of subjects implanted with a Lotus Valve). Reported as percent of subjects.
Effective orifice area | At discharge from hospital or at 7 days post-procedure (whichever comes first)
  Effective orifice area as measured by echocardiography and assessed by an independent core laboratory
Successful repositioning of the study valve if repositioning is attempted | Immediately post-procedure (patient discharged from operative room)
Successful retrieval of the study valve if retrieval is attempted | Immediately post-procedure (patient discharged from operative room)
Grade of paravalvular aortic regurgitation | At discharge from hospital or at 7 days post-procedure (whichever comes first)
  Grade of paravalvular aortic regurgitation as measured by echocardiography and assessed by an independent core laboratory

OTHER OUTCOMES:
Mortality: all-cause, cardiovascular, and non-cardiovascular | At discharge or 7 days post-procedure (whichever comes first), 30 days, 6 months, and 1 year post procedure
Stroke: disabling and non-disabling | At discharge or 7 days post-procedure (whichever comes first), 30 days, 6 months, and 1 year post procedure
Myocardial infarction (MI): periprocedural (≤72 hours post index procedure) and spontaneous (>72 hours post index procedure) | At discharge or 7 days post-procedure (whichever comes first), 30 days, 6 months, and 1 year post procedure
Bleeding: life-threatening (or disabling) and major | At discharge or 7 days post-procedure (whichever comes first), 30 days, 6 months, and 1 year post procedure
Acute kidney injury based on the AKIN System Stage 3 (including renal replacement therapy) or Stage 2 | At discharge or 7 days post-procedure (whichever comes first), 30 days, 6 months, and 1 year post procedure
Major vascular complication | At discharge or 7 days post-procedure (whichever comes first), 30 days, 6 months, and 1 year post procedure
Repeat procedure for valve-related dysfunction (surgical or interventional therapy) | At discharge or 7 days post-procedure (whichever comes first), 30 days, 6 months, and 1 year post procedure
Hospitalization for valve-related symptoms or worsening congestive heart failure (New York Hear Association [NYHA] class III or IV) | At discharge or 7 days post-procedure (whichever comes first), 30 days, 6 months, and 1 year post procedure
New permanent pacemaker implantation resulting from new or worsened conduction disturbances (including new left bundle branch block [LBBB] and third degree atrioventricular block) | At discharge or 7 days post-procedure (whichever comes first), 30 days, 6 months, and 1 year post procedure
New onset of atrial fibrillation or atrial flutter | At discharge or 7 days post-procedure (whichever comes first), 30 days, 6 months, and 1 year post procedure
Coronary obstruction | ≤72 hours post index procedure
Ventricular septal perforation | ≤72 hours post index procedure
Mitral apparatus damage | ≤72 hours post index procedure
Cardiac tamponade | ≤72 hours post index procedure
Prosthetic aortic valve malpositioning, including valve migration, valve embolization, or ectopic valve deployment | At discharge or 7 days post-procedure (whichever comes first), 30 days, 6 months, and 1 year post procedure
Transcatheter aortic valve (TAV)-in-TAV deployment | At discharge or 7 days post-procedure (whichever comes first), 30 days, 6 months, and 1 year post procedure
Prosthetic aortic valve thrombosis | At discharge or 7 days post-procedure (whichever comes first), 30 days, 6 months, and 1 year post procedure
Prosthetic aortic valve endocarditis | At discharge or 7 days post-procedure (whichever comes first), 30 days, 6 months, and 1 year post procedure
Prosthetic aortic valve performance: effective orifice area | 30 days, 6 months, and 1 year post procedure
  Measured by transthoracic echocardiography (TTE) and assessed by an independent core laboratory
Prosthetic aortic valve performance: mean pressure gradient | 30 days, 6 months, and 1 year post procedure
  Measured by transthoracic echocardiography (TTE) and assessed by an independent core laboratory
Prosthetic aortic valve performance: aortic valve regurgitation | At discharge or 7 days post-procedure (whichever comes first), 30 days, 6 months, and 1 year post procedure
  Measured by transthoracic echocardiography (TTE) and assessed by an independent core laboratory
Prosthetic aortic valve performance: peak gradient | At discharge or 7 days post-procedure (whichever comes first), 30 days, 6 months, and 1 year post procedure
  Measured by transthoracic echocardiography (TTE) and assessed by an independent core laboratory
Prosthetic aortic valve performance: peak velocity | At discharge or 7 days post-procedure (whichever comes first), 30 days, 6 months, and 1 year post procedure
  Measured by transthoracic echocardiography (TTE) and assessed by an independent core laboratory
Functional status as evaluated by New York Heart Association (NYHA) classification | At discharge or 7 days post-procedure (whichever comes first), 30 days, 6 months, and 1 year post procedure
Neurological status: National Institutes of Health Stroke Scale (NIHSS) | At discharge and 1 year
Neurological status: Modified Rankin Scale (mRS) | At discharge or 7 days post-procedure (whichever comes first), 30 days, 6 months, and 1 year post procedure

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Götberg, MD, PhD, Principal Investigator — Skane University Hospital; Sabine Bleiziffer, MD, Principal Investigator — German Heart Centre München
Locations (3):
- Rigshospitalet, Copenhagen, Denmark
- Clinique Pasteur, Toulouse, France
- Skåne University Hospital, Lund, Sweden

IPD SHARING:
Plan to Share IPD: No